CLINICAL TRIAL: NCT03301805
Title: A Phase II, Open Label Study to Evaluate the Safety and Efficacy of BLEX 404 Oral Liquid Combined With Gemcitabine Monotherapy in Patients With Advanced Inoperable or Metastatic Pancreatic Cancer
Brief Title: A Phase II, EvaluateBLEX 404 Combined With Gemcitabine Monotherapy With Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rgene Corporation (Industry)
Collaborators: American BriVision Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGC-1502-01
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Study Objectives Part I To determine the safety and recommended dose level (RDL) of BLEX 404 Oral Liquid combined with Gemcitabine monotherapy in a 28-day schedule.
  Part II To assess the efficacy and safety of BLEX 404 Oral Liquid combined with Gemcitabine monotherapy at the recommended dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BLEX 404 Oral Liquid (Experimental): During Phase I study (dose escalation), a standard 3+3 design will be followed, and the dose range is 3 to 10 mg/kg BID. The recommended dose level (RDL) for the Phase II study is defined as the dose level with 0 to 1 DLT observed during cycle I of Gemcitabine monotherapy among 6 patients in the Phase I study.
  Interventions: Drug: BLEX 404

INTERVENTIONS:
Drug: BLEX 404 — BLEX 404 Oral Liquid is administered twice daily during the Gemcitabine monotherapy period. The dose of Gemcitabine 1,000 mg/m2 IV fusion at Day 1, 8, 15 of every cycle
  * 28 days a cycle.

SUMMARY:
The primary purpose of this study is to determine the safety and recommended dose level (RDL) of BLEX 404 Oral Liquid combined with Gemcitabine monotherapy in a 28-day schedule.The secondary purpose is to assess the efficacy and safety of BLEX 404 Oral Liquid combined with Gemcitabine monotherapy at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 - 80 years old at the time of signing the ICF.
2. Patients with pathologically proved adenocarcinoma of pancreatic cancer and diagnosed with inoperable/metastatic disease (previous systemic chemotherapy, neoadjuvant or adjuvant gemcitabine are acceptable, unless exclusion criteria met).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 1 to 2.
4. Adequate hematologic function defined as: absolute neutrophil count (ANC) >= 2,000/μL; platelets count >= 100,000/μL; hemoglobin must be >= 10 g/dL (can be corrected by growth factor or transfusion).
5. Adequate hepatic function defined as: serum bilirubin =< 1.5-fold upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 3-fold ULN (5-fold ULN if liver metastasis is observed).
6. Adequate renal function with: serum creatinine =< 1.3 mg/dL or calculated creatinine clearance >= 60 mL/minute according to the Cockcroft and Gault formula.
7. At least one measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
8. Women must be either of non-child bearing potential, or women with child-bearing potential agree to use effective a highly contraceptive method or a contraceptive implant, exception of hormonal contraception (estrogen/progesterone), during treatment from time of Screening Visit and after cessation of therapy at least 3 months.
9. Planning to receive Gemcitabine monotherapy.
10. Willing and able to comply with all aspects of the treatment protocol.
11. Provide written informed consent.

Exclusion Criteria:

1. Patients with following treatment prior to Gemcitabine monotherapy: chemotherapy, immunotherapy, or biologic systemic anticancer therapy within 28 days of study entry.
2. Pancreatic patients with prior history of Gemcitabine chemotherapy.
3. Women who are pregnant or breastfeeding.
4. Patients with brain metastasis.
5. Patients with bone metastasis alone.
6. Patients with autoimmune disease that requires systemic steroids or immunosuppression agents.
7. Current enrollment in another clinical study or used any investigational drug or device within the past 28 days preceding informed consent.
8. Known history of human immunodeficiency virus (HIV) infection.
9. Existing anticancer treatment-related toxicities of Grades >= 2 (except for alopecia and neuropathy) according to Common Terminology Criteria for Adverse Events (CTCAE v4.03).
10. Patients with an active infection requiring systemic therapy.
11. Patients are hepatitis C virus (HCV) carrier, and/or with active viral disease which is defined as hepatitis B virus (HBV) carrier with HBV DNA > 2,000 IU/ml plus AST and ALT > 3-fold ULN.
12. History of concomitant medical conditions or infectious diseases that, in the opinion of the investigator, would compromise the patient's ability to safely complete the study.
13. Ascertained hypersensitivity to investigational product, Gemcitabine or any of the excipients used in the study.
14. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily BLEX 404 Oral Liquid treatment.
15. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation, psychiatric disorder, with any other serious diseases/medical history.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Part I: Dose-limiting toxicity (DLT) observation | 4 weeks (1 cycle)
  Presence or absence of dose-limiting toxicity (DLT) related to BLEX 404 Oral Liquid for each patient during first cycle of Gemcitabine monotherapy to determine the recommended dose level (RDL).
Part II: Overall response rate (PR + CR) | 12 weeks (3 cycle)
  Overall response rate (PR + CR) after 4 cycles of combination use in BLEX 404 + Gemcitabine monotherapy.

SECONDARY OUTCOMES:
Part II: Overall benefit rate (CR + PR + SD) | 12 weeks (3 cycle)
  1. Overall benefit rate (CR + PR + SD) after at least 3 cycles of combination use of BLEX 404 plus Gemcitabine monotherapy.
Part II: Incidence of grade 3/4 hematological toxicity | 4 weeks (1 cycle)
  Rate of grade 3/4 hematological toxicity of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Gi-Ming Lai, M.D., Principal Investigator — Taipei Municipal Wanfang Hospital

IPD SHARING:
Plan to Share IPD: No